CLINICAL TRIAL: NCT03629678
Title: Using Patient-Centered Guidelines in a Technology Platform to Improve Health Care in Adults With Sickle Cell Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: Ohio State University (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Robert M Cronin, MD, MS, Assistant Professor, Vanderbilt University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K23HL141447-2; K23HL141447 (NIH)
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Results first posted 2024-06-27 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Sickle Cell Disease
Keywords: mhealth
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Booklets) (No Intervention): Group 1 will receive the control arm with a paper booklet of the patient-centered SCD-guidelines with education by a health care provider at a single visit
- mobile health application (Active Comparator): Group 2 will receive continuous access to technology-based patient-centered SCD-specific guidelines using a user-driven technological platform, plus a paper booklet of the guidelines with education by a health care provider at a single visit. The mobile app will include interactive content and a fully searchable collection of the SCD-specific guidelines that are age- and health literacy-appropriate. Through the mobile app, the investigators will reinforce important points of guideline content; motivate patient engagement through quizzes and reminders; and facilitate peer support, for instance by forming teams to compete against each other to attain goals.
  Interventions: Other: mobile health application

INTERVENTIONS:
Other: mobile health application — The user-driven technological tool will include an mHealth mobile phone application. Features of the application will be based on preliminary work from the investigators' sites. The mobile app will include fully searchable provider-facing and patient-facing interfaces with the SCD-specific guidelines. The provider-facing interface, designed to be used by providers, will be separated by patient's age to accommodate pediatric and adult providers. The patient-facing interface will display the guidelines that are age- and health literacy-appropriate. Through the mobile app, the investigators will reinforce important points of guideline content; motivate patient engagement through quizzes and text-message reminders; and facilitate peer support, for instance by forming teams to compete against each other to attain goals.
  Arms: mobile health application

SUMMARY:
SCD is an inherited disorder of hemoglobin that affects over 100,000 Americans, most of whom live in low-resourced neighborhoods. Acute SCD complications result in 230,000 emergency department visits and $1.5 billion annually in acute-care expenditures. Prior research indicates that increased disease-specific knowledge correlates with improved clinical outcomes in SCD. Thus, targeting strategies to improve disease-specific knowledge is a high priority in the care of individuals with SCD. Significant evidence describes how educational materials, including online educational programs, can be used to increase disease-specific knowledge. In this study, the investigators will evaluate a mobile phone technology intervention based on the prior evidence that technologies can improve SCD-specific knowledge.

DETAILED DESCRIPTION:
Sickle cell disease (SCD) is an inherited blood disorder that affects over 100,000 Americans, an underserved population with low life expectancy and risk for significant and life-threatening medical complications (e.g., stroke). Adults with SCD are overwhelmingly members of socially disadvantaged groups, increasing their risk for disparities in care. Annual health expenditure for individuals with SCD in the United States is about $1.5 billion, primarily from multiple emergency room visits (230,000 visits/year) for management of acute complications. Use of disease-specific knowledge has emerged as a powerful tool to decrease health care utilization. Significant evidence has described how to increase disease-specific knowledge using educational materials, including online educational programs in individuals managing chronic diseases, including SCD. Patient knowledge and use of disease-specific information like evidence-based clinical guidelines has the potential to decrease health care utilization. In 2014, the National Heart, Lung, and Blood Institute (NHLBI) published guidelines for evidence-based management of SCD for health care providers. However, to date, no national strategy has been developed to make these guidelines patient-centered, accessible, and actionable for adults with SCD. Federal Meaningful Use regulations have recommended using health-related technologies to improve patient access to their health information to promote patient engagement. Yet, many adults with SCD are not yet fully engaged in use of health technologies because they are unsure of the best format (e.g., mobile or web-based), leading to a health care technology gap. Mobile health applications (apps) that include patient-centered care guidelines could engage and activate this population given the high use of mobile technologies, potentially closing this health technology gap and improving health outcomes.

Evaluate the feasibility and acceptability of the refined iManage in a pilot study with adults with SCD. The investigators will recruit 50 adults from the population of 250 adults with SCD at the Vanderbilt Meharry Sickle Cell Disease Center of Excellence and the ohio state university comprehensive sickle cell center for a 6-month pilot study to evaluate usability, acceptance, and usage. At the end of the study, the investigators will conduct interviews with a subset of participants to gain an in-depth understanding of usage patterns and how to sustain engagement to promote ongoing app use.

Evaluate the efficacy of the refined iManage app on SCD-specific knowledge. The investigators will test the hypothesis that the refined iManage will increase SCD-specific knowledge by measuring SCD-specific knowledge at the start and end of the 6-month pilot study. the investigators will conduct exploratory analyses of secondary outcomes including patient activation, adherence to guidelines, missed days of school/work, and self-efficacy.

ELIGIBILITY:
Inclusion Criteria:

* receives care at the community health clinic,
* diagnosis of SCD (Hgb SS, SC, Sβ-thal),
* ability to speak and understand written English
* has access to a smartphone or computer
* between 18-70 years.

Exclusion Criteria:

* lack of access to a smartphone or computer
* inability to speak and understand written English

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Ohio State University Medical Center, Columbus, Ohio
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Cronin RM, Quaye N, Liu X, Landes K, Crosby LE, Kassim AA, Volanakis EJ, Schnell PM, DeBaun MR. A feasibility randomized controlled trial of an mHealth app vs booklets for patient-facing guidelines in adults with SCD. Blood Adv. 2023 Oct 24;7(20):6184-6190. doi: 10.1182/bloodadvances.2023010676. PMID 37595029

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We conducted a feasibility randomized controlled trial at two centers: Vanderbilt University Medical Center and the Ohio State University, between 2018-2022. The IRBs approved the trial at each institution. Participants were recruited from sickle cell medical clinics.
Groups:
- Mobile Health Application: Group 2 will receive continuous access to technology-based patient-centered SCD-specific guidelines using a user-driven technological platform, plus a paper booklet of the guidelines with education by a health care provider at a single visit. The mobile app will include interactive content and a fully searchable collection of the SCD-specific guidelines that are age- and health literacy-appropriate. Through the mobile app, the investigators will reinforce important points of guideline content; motivate patient engagement.
  mobile health application: The user-driven technological tool will include an mHealth mobile phone application. Features of the application will be based on preliminary work from the investigators' sites. The mobile app will include fully searchable provider-facing and patient-facing interfaces with the SCD-specific guidelines. The provider-facing interface, designed to be used by providers, will be separated by patient's age to accommodate pediatric and adult providers. The patient-facing interface will display the guidelines that are age- and health literacy-appropriate. Through the mobile app, the investigators will reinforce important points of guideline content; motivate patient engagement through quizzes and text-message reminders; and facilitate peer support, for instance by forming teams to compete against each other to attain goals.
Period: Overall Study
Arm/Group | Control Group (Booklets) | Mobile Health Application
Started | 30 | 37
Completed | 25 | 31
Not Completed | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Mobile Health Application: Group 2 will receive continuous access to technology-based patient-centered SCD-specific guidelines using a user-driven technological platform, plus a paper booklet of the guidelines with education by a health care provider at a single visit. The mobile app will include interactive content and a fully searchable collection of the SCD-specific guidelines that are age- and health literacy-appropriate.
  mobile health application: The user-driven technological tool will include an mHealth mobile phone application. Features of the application will be based on preliminary work from the investigators' sites. The mobile app will include fully searchable provider-facing and patient-facing interfaces with the SCD-specific guidelines. The provider-facing interface, designed to be used by providers, will be separated by patient's age to accommodate pediatric and adult providers. The patient-facing interface will display the guidelines that are age- and health literacy-appropriate. Through the mobile app, the investigators will reinforce important points of guideline content; motivate patient engagement through quizzes and text-message reminders; and facilitate peer support, for instance by forming teams to compete against each other to attain goals.
- Total: Total of all reporting groups
Arm/Group | Control Group (Booklets) | Mobile Health Application | Total
Number analyzed (Participants) | 25 | 31 | 56
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 25 | 30 | 55
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (8.82) | 35.6 (10.9) | 33.5 (10.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 16 | 25
  Male | 16 | 15 | 31
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 24 | 27 | 51
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 23 | 31 | 54
  White | 0 | 0 | 0
  More than one race | 2 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 25 | 31 | 56
Sickle cell genotype [Count of Participants; unit: Participants]
  Hemoglobin SS / Sbeta0 thalassemia | 14 | 19 | 33
  Hemoglobin SC / Sbeta+ thalassemia | 10 | 12 | 22
  Don't know | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: SCD-specific Knowledge
Description: Knowledge about SCD. This is a questionnaire that is multiple choice and asks questions about sickle cell disease with one correct answer and 3 incorrect answers. The investigators will sum up the number of correct answers which will be reported. There were a total of 39 questions, so a maximum score of 39.
  This is not a scale.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group (Booklets) | Mobile Health Application
Number analyzed (Participants) | 24 | 26
score on a scale
  Baseline | 32.0 [12.0 to 37.0] | 32.0 [18.0 to 37.0]
  6-month follow up | 33.5 [16 to 37] | 33 [22 to 39]

2. Secondary Outcome: Self-efficacy
Description: sickle cell self-efficacy scale, as described in Edwards R, Telfair J, Cecil H, Lenoci J. Reliability and validity of a self-efficacy instrument specific to sickle cell disease. Behav Res Ther. 2000;38(9):951-63.
  Scale is 0-45, higher score is better Scale has no subscales and measures self-efficacy
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Groups:
- Mobile Health Application: Group 2 will receive continuous access to technology-based patient-centered SCD-specific guidelines using a user-driven technological platform, plus a paper booklet of the guidelines with education by a health care provider at a single visit. The mobile app will include interactive content and a fully searchable collection of the SCD-specific guidelines that are age- and health literacy-appropriate. Through the mobile app, the investigators will reinforce important points of guideline content; motivate patient engagement through quizzes and reminders; and facilitate peer support.
  mobile health application: The user-driven technological tool will include an mHealth mobile phone application. Features of the application will be based on preliminary work from the investigators' sites. The mobile app will include fully searchable provider-facing and patient-facing interfaces with the SCD-specific guidelines. The provider-facing interface, designed to be used by providers, will be separated by patient's age to accommodate pediatric and adult providers. The patient-facing interface will display the guidelines that are age- and health literacy-appropriate. Through the mobile app, the investigators will reinforce important points of guideline content; motivate patient engagement through quizzes and text-message reminders; and facilitate peer support, for instance by forming teams to compete against each other to attain goals.
Arm/Group | Control Group (Booklets) | Mobile Health Application
Number analyzed (Participants) | 24 | 26
score on a scale | 34.5 [27 to 37] | 32.5 [27.2 to 36]

3. Secondary Outcome: Healthcare Utilization (ER Visits and Hospitalizations)
Description: The investigators will measure a count of the # ER visits and # of hospitalizations (i.e., # ER visits + # hospitalizations)
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: events
Arm/Group | Control Group (Booklets) | Mobile Health Application
Number analyzed (Participants) | 24 | 26
events | 0 [0 to 1] | 0 [0 to 0]

4. Secondary Outcome: Usage and Usability of the mHealth Application
Description: How often app and functionality was used. Usability will be measured by the widely used and validated System Usability Scale as described in Brooke J. SUS-A quick and dirty usability scale. Usability evaluation in industry. 1996;189(194):4-7. The mobile health application for the guidelines has built-in tracking of the number of times the application is launched, how many times each of the functions are used, and how many times each button has been pushed. To measure usage, the investigators will record the numbers of each of these events for each participant. In addition to total use, the investigators will measure usage over time including any use, initial use, periodic use, and sustained use.
  SUS scale is 0-100, higher score is better. Scale has no subscales and measures usability of the app
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Mobile Health Application
Number analyzed (Participants) | 26
score on a scale | 56.2 [50 to 68.8]

5. Secondary Outcome: Patient Activation Measure
Description: The Patient Activation Measure (PAM) is a 10-item questionnaire to assesses a patient's knowledge, skills, and confidence in managing their health and healthcare. Response options range from (1) disagree strongly to (4) agree strongly, and an additional "not applicable" option. The sum of responses (excepting non-applicable items) are converted using Insignia Health's proprietary algorithm (that takes into account the specific wording and weighting of each item in the survey) into a final PAM score on a 0-100 scale. Higher PAM scores indicate a greater level of patient activation in managing their health.
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Control Group (Booklets) | Mobile Health Application
Number analyzed (Participants) | 24 | 26
score on a scale | 73.8 [58.5 to 100] | 73.8 [56 to 85.3]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Control Group (Booklets) | Mobile Health Application
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/37
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/37
Other Adverse Events (participants affected / at risk) | 0/30 | 0/37

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-20): https://cdn.clinicaltrials.gov/large-docs/78/NCT03629678/Prot_SAP_000.pdf